CLINICAL TRIAL: NCT02475863
Title: A Study to Compare Model-based Warfarin Dosing to the Traditional Approach in Children After Congenital Heart Surgery at Glenfield Hospital, Leicester
Brief Title: Model-based Versus Traditional Warfarin Dosing in Children
Acronym: WATCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: De Montfort University (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: DMU-1527
Record Dates: First submitted 2015-06-12; First posted 2015-06-19 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Congenital Heart Defects
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Warfarin dosing aid (Experimental): A pharmacokinetic/pharmacodynamic model-based dosing algorithm for warfarin.
  Interventions: Device: Warfarin Dosing Aid
- Standard practice (Active Comparator): Dosing adjustments according to the normal unit protocol
  Interventions: Other: Standard Practice

INTERVENTIONS:
Device: Warfarin Dosing Aid — A pharmacokinetic/pharmacodynamic model-based dosing algorithm for warfarin
  Arms: Warfarin dosing aid
Other: Standard Practice — Warfarin dose adjustments according to standard unit protocol
  Arms: Standard practice

SUMMARY:
This study compares the clinical effectiveness of a new algorithm (model-based warfarin dosing) with standard practice (doctor's own judgement and intuition) designed to determine the most appropriate anticoagulant dose of warfarin in children after congenital heart surgery.

DETAILED DESCRIPTION:
Warfarin is widely used in children after heart surgery in order to prevent complications that may arise due to blood clots forming in unwanted places - for example in the brain causing a stroke. If too little warfarin is given, there is a risk that clots may form. If the dose is too high, bleeding will result.

Traditionally, the approach to dosing warfarin in children has been to select a starting dose according to standard guidelines and to then adjust the doses for each child by monitoring the INR (which measures how quickly blood clots). However, a person's make up as well as external factors, such as age, weight, diet and genetics can affect warfarin dosing and this makes controlling the dose and hence controlling the INR, more difficult. Recently however, a more sophisticated dosing model has been developed by researchers which takes into account some of these factors. The model is designed to help doctors select the best dose of warfarin for children by individualising prescriptions.

The aim of the proposed research is, therefore, to compare the model based warfarin dosing with the traditional approach to warfarin dosing in children who have undergone congenital heart surgery. The research will involve children who are started on warfarin for the first time and also children who are already receiving ongoing warfarin therapy.

ELIGIBILITY:
Inclusion Criteria: -Children from birth up to 18 years with congenital heart disease who have been treated or to be treated with warfarin after undergoing reconstructive heart surgery at Glenfield Hospital, Leicester, United Kingdom.

Exclusion Criteria:

1. Patients aged over 18 years who are treated as 'adults'.
2. Children who refuse assent, parents who refuse consent.
3. Any significant disease or disorder which, in the opinion of the direct care team, may either put the participant at risk because of study participation or adversely affect the participants' ability to participate in the study.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
The difference between the model based and traditional warfarin dosing method in International Normalised Ratio (INR) response. | 6 months for warfarin naiive patients and 12 months for patients already on warfarin therapy.
  INR response includes: Time taken (days per patient) to achieve stable anticoagulation within the desired therapeutic range (TR), number and percentage of INR measurements within the TR, Time in TR, and frequency of INR measurements (number of INR measurements per month) per patient.

SECONDARY OUTCOMES:
Medical staff perceptions of value of warfarin dosing aid | Within six months of end of period of data collection
  Interviews with medical staff will be conducted
Patients or carers 'lived experience' of monitoring warfarin dosing and INR | Within six months of end of cross-over trial
  Interviews will be conducted with patients and or carers
The incidence of warfarin-related adverse events, bleeding and bruising, by recording on symptom diary cards | 6 months for warfarin naiive patients and 12 months for patients already on warfarin therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hussain Mulla, PhD, Principal Investigator — Univesity Hospitals Leicester NHS Trust